CLINICAL TRIAL: NCT06090435
Title: Movement Simulation Techniques and Therapeutic Exercise in Young Nulliparous Women: A Randomized Controlled Trial
Brief Title: Movement Simulation Techniques and Therapeutic Exercise in Young Nulliparous Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ferran Cuenca, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV0002
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Motor Imagery; Action Observation; Therapeutic Exercise
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic exercise plus motor imagery (Experimental)
  Interventions: Behavioral: Therapeutic exercise plus motor imagery
- Therapeutic exercise plus action observation (Experimental)
  Interventions: Behavioral: Therapeutic exercise plus action observation
- Therapeutic exercise (Active Comparator)
  Interventions: Behavioral: Therapeutic exercise

INTERVENTIONS:
Behavioral: Therapeutic exercise plus motor imagery — Therapeutic exercise programme (aerobic exercise and strengthening exercise) to which is added a motor imagery intervention (which consists of imagining the same movements but not performing them for real).
  Arms: Therapeutic exercise plus motor imagery
Behavioral: Therapeutic exercise plus action observation — Therapeutic exercise programme (aerobic exercise and strengthening exercise) to which is added an action observation intervention (which consists of observing the same movements but not performing them for real).
  Arms: Therapeutic exercise plus action observation
Behavioral: Therapeutic exercise — Therapeutic exercise programme (aerobic exercise and strengthening exercise) to which is added a sham action observation intervention (which consists of observing planets in space).
  Arms: Therapeutic exercise

SUMMARY:
Both motor imagery and action observation training, either alone or in combination with physical practice, have been shown to improve some clinical variables of interest such as strength and motor control. However, this has not yet been investigated in the pelvic floor musculature.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and asymptomatic women.

Exclusion Criteria:

* This study will exclude those who presented a respiratory pathology, cardiac, systematic, or metabolic disease, history of recent surgery, vertebral fracture, or osteoarticular disorders of the spine area.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
maximal pelvic floor muscle strength (measured in grams and with the phenix device) | pre-intervention (T0), at one week after the intervention (T1) and at two weeks after starting the intervention (post-intervention (T2)).
  Three measurements of maximal pelvic floor strength shall be performed with an intracavitary probe and the mean of the three measurements of maximal pelvic floor muscle strength shall be considered.
Algometry for assessing pressure pain thresholds (Pain sensitivity) | pre-intervention (T0), at one week after the intervention (T1) and at two weeks after starting the intervention (post-intervention (T2)).
  An algometer shall be used to assess pain thresholds to pressure, i.e. squeezing so that pressure is converted into pain at four points. Two points in the symphysis pubis area, one point in the lumbar area and one point near the tibial tuberosity.
Motor control of the lumbopelvic area assessed with a biofeedback device. | pre-intervention (T0), at one week after the intervention (T1) and at two weeks after starting the intervention (post-intervention (T2)).
  A protocol to assess lumbopelvic dissociation (i.e. moving the legs without moving the lower back) of both legs of the participants will be performed with a biofeedback device that assesses the pressure exerted on the lower back during leg mobilisation (in mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Ferran Cuenca Martínez, Valencia, Spain